CLINICAL TRIAL: NCT01712893
Title: A Phase III,Randomized,Open Label Study Comparing Simultaneous Versus Sequential Use of Adjuvant Chemotherapy and GnRHa up to 2-3 Years for ≤ 45 Year Old Pre-menopausal Hormone Receptor-positive Breast Cancer
Brief Title: Simultaneous Versus Sequential Use of Adjuvant Chemotherapy and GnRHa in Treating ER+,Premenopausal Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of Department of Surgical Oncology,Cancer Hospital & Institute, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD trial
Record Dates: First submitted 2012-10-21; First posted 2012-10-24 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant therapy; Ovarian suppression
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoladex combined with chemotherapy (Experimental): After signing informed consent, patients will be screened, eligible patients were randomly divided into 2 groups, the test group should use Zoladex 3.6mg once a month up to 2-3 years combined with chemotherapy,all patients will receive Tamoxifen after chemotherapy
  Interventions: Drug: Zoladex
- Zoladex after chemotherapy (Active Comparator): After signing informed consent, patients will be screened, eligible patients were randomly divided into 2 groups, the control group should use Zoladex 3.6mg once a month up to 2-3 years after chemotherapy,all patients will receive Tamoxifen after chemotherapy
  Interventions: Drug: Zoladex

INTERVENTIONS:
Drug: Zoladex — Eligible patients were randomly divided into 2 groups, the intervention group should use Zoladex 3.6mg once a month up to 2-3 years combined with chemotherapy,and the control group should use chemotherapy alone followed by Zoladex
  Other Names: Zoladex = GnRHa,Goserelin

SUMMARY:
The present study is a randomized open-label -phase III study that aims to compare the efficacy and safety of the adjuvant chemotherapy with simultaneous or sequential application of Zoladex up to 2-3 years for ≤ 45 year old premenopausal hormone receptor-positive breast cancer.

DETAILED DESCRIPTION:
Data showed that ovarian suppression therapy may protect the ovarian function in premenopausal patients received chemotherapy for breast cancer. However this is still a controversial issue. Sequential use of GnRHa (Zoladex) as ovarian suppression treatment after chemotherapy has been established as an effective endocrine therapy for ER positive premenopausal breast cancer. The present study is a randomized open-label phase III study that aims to observe the efficacy and safety of the adjuvant chemotherapy with simultaneous combination of Zoladex up to 2-3years and chemotherapy compared with the sequential schedule in ≤ 45 year old premenopausal hormone receptor-positive breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. female
2. Primary invasive breast cancer pathologically approved by core needle or open biopsy
3. Patients must have undergone standard surgery for primary breast cancer as shown in the following:

   * mastectomy
   * breast conservation surgery followed by whole breast radiation
   * axillary dissection or sentinel node biopsy
4. Need adjuvant chemotherapy after surgery
5. Patients taking neo-chemotherapy are eligible
6. Patients with synchronous bilateral cancers are eligible on the condition that If one side is IDC and the other side is DCIS, the IDC side should be of the ER and/or PR positive phenotype and IF two sides are both IDC, they must be ER and/or PR positive phenotype at the same time
7. Hormone receptor positive (≥＋) is defined as detecting ER or PR expression at any time is eligible. The situation of only PR positive and ER negative is eligible, too
8. Based on the study objective, all patients are required to be premenopausal as defined by

   * menstruating actively
   * less than 6 months since last menstrual period (LMP), or patients younger than 40 years of age who became amenorrheic not more than 1 year if the serum free E2、FSH and LH level was premenopausal (according to the reference value of local center).
   * had previous hysterectomy with one or both ovaries left intact are eligible if the serum free E2、FSH and LH level are premenopausal (according to the reference value of local center).
9. patients must have an ECOG performance status of 0 or 1 (0-fully active, able to carry on all pre-disease performance without restriction, 1-restricted in physical strenuous actively but ambulatory)
10. leucocyte count must be ≥ 3.0*10^9/L and platelet count must be ≥ 100*10^9/L
11. AST/SGOT or ALT/AGPT must be < 3 times the ULN
12. serum creatinine must be < 2 times the ULN
13. pregnancy testing is negative and are willing to do contraception during the treatment period

Exclusion Criteria:

1. patients with metastatic malignant tumor
2. previous history of asynchronous bilateral breast cancer
3. any previous malignancy in the past 5 years, except for those treated with curative intent, such as carcinoma in situ of the cervix, squamous carcinoma of the skin or basal cell carcinoma of the skin
4. any non-malignant systemic disease which interfere long time follow up
5. history of medical ovarian ablation therapy
6. severe live dysfunction, Child-Pugh is grade C
7. Severe renal dysfunction
8. Occult breast cancer
9. severe heart dysfunction, heart functional classification is above Class III

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2009-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Resumption of menstruation | 1 year
  the Resumption that patients recover the natural menstrual or serum E2, FSH, LH return to the premenopausal range within 1 year after stopping Zoladex

SECONDARY OUTCOMES:
RFS | 5years
  Relapse free survival (RFS): RFS related events ware defined as local-regional recurrence, distant metastasis or death, whichever occurred first.during follow up
OS | 5 years
  Overall survival
Other adverse events | 5years
  Other adverse events (Gynecological events, blood lipids, thrombosis, cardiovascular diseases, and etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Min Shao, MD, Principal Investigator — Fudan University
Locations (1):
- FUSCC, Shanghai, Shanghai Municipality, China